CLINICAL TRIAL: NCT03933397
Title: A Comparison of Individualized vs. Weight Based Protocols to Treat Vaso-Occlusive Episodes in Sickle Cell Disease
Brief Title: Comparing Individualized vs. Weight Based Protocols to Treat Vaso-Occlusive Episodes in Sickle Cell Disease
Acronym: COMPARE-VOE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to COVID enrollment numbers needed to meet the primary endpoint will not be met.
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00101245; 1U24HL137907-01A1 (NIH)
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Morphine; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient-Specific Protocol (Experimental): Patients assigned to this treatment protocol will be given pain medicine(s) based on the pain medicine(s) they take at home, what was needed during their past hospital and emergency department visits to treat pain and doses that have been effective and safe in the past.
  Interventions: Other: Patient-Specific Protocol; Drug: Morphine; Drug: Hydromorphone
- Weight-based Protocol (Experimental): Patients assigned to this treatment protocol will be given pain medicine(s) based on their weight.
  Interventions: Other: Weight-based Protocol; Drug: Morphine; Drug: Hydromorphone

INTERVENTIONS:
Other: Patient-Specific Protocol — Patients assigned to this treatment protocol will be given pain medicine(s) based on the pain medicine(s) they take at home for pain and what was needed during their past hospital and emergency department visits to treat pain. Medicines will include opioids, either morphine or hydromorphone. A member of the outpatient SCD provider team will review the patient's medical record to determine: 1) the patient's maximum home opioid dose, and 2) previous ED analgesic medication(s) and doses that have been effective and safe in the past. The patient's regular hematologist/sickle cell team will write the treatment plans. Medications will be given every 20-30 minutes for up to 6 hours.
  Arms: Patient-Specific Protocol
Other: Weight-based Protocol — Patients assigned to this treatment protocol will be given pain medicine(s) based on their weight. Medicines will include opioids, either morphine or hydromorphone. Plans will be written by the patients regular hematologist/sickle cell team.
  Arms: Weight-based Protocol
Drug: Morphine — 4 mg for participants weighing <50 kgs, 6mg for participants weighing 50-69.9 kgs, 8mg for participants weighing 70 - 89.9 kgs and 10mg for participants weighing greater than or equal to 90 kgs. dose is given. Re-dosing is every 20-30 minutes up to 6 hours with one possible dose escalation of 25%.
  Other Names: Morphine Sulfate
Drug: Hydromorphone — 1 mg for participants weighing <60 kgs, 1.5 mg for participants weighing 60 - 89.9 kgs, and 2 mg for participants weighing greater than or equal to 90 kgs. dose is given. Re-dosing is every 20-30 minutes up to 6 hours with one possible dose escalation of 25%.
  Other Names: Dilaudid

SUMMARY:
The purpose of this research study is to compare two different ways to give opioid pain medicine to treat sickle cell disease pain that is bad enough to go to the emergency department for treatment. One way uses your weight to decide how much pain medicine to give you while in the emergency department. This is called weight based treatment. The other way uses how much pain medicine you take at home and how much medicine you needed during past emergency department visits to decide how much medicine to give you. This is called patient specific treatment.

ELIGIBILITY:
Inclusion Criteria:

* All adult (18 years or older);
* Sickle Cell Disease patients with the following genotypes: Hgb SS (sickle cell anemia), SC(Sickle hemoglobin-c) , and SB+(sickle Beta-Plus thalassemia) and SB-(sickle Beta zero thalassemia)

Exclusion Criteria:

* determined to not benefit from opioids and therefore won't receive opioids in any future Emergency Department visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huiman Barnhart, PhD, Principal Investigator — Duke University; Paula Tanabe, PhD, Principal Investigator — Duke University School of Nursing
Locations (6):
- United States (6):
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - Atrium Health, Charlotte, North Carolina
  - Case Western University, Cleveland, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between August 13, 2019 - May 13 2022 at 6 academic institutions. Institutions selected based on minimum average of two ED (Emergency Department) visits/day by patients with SCD(Sickle Cell Disease) for treatment of VOE (Vaso-occlusive pain events), hematologist willing to randomize patients to the treatment arms, informatics support to post the protocols in electronic health record and infrastructure to support both enrollment of subjects and prospective data collection.
Pre-assignment Details: Participants were consented & randomized in ED, clinic or by phone with the onset of COVID-19. Pain protocols were written based on the randomization arm assigned and uploaded to the Electronic Medical Record for use if the participant presented to the emergency department (ED) for pain related to their sickle cell disease. Patients were evaluated for COVID-19 at the ED visit & excluded if COVID positive. During the ED visit, baseline date were collected following bed placement of participant.
Groups:
- Patient-Specific Protocol: Patients assigned to this arm will be given pain medicine(s) based on pain medicine(s) they take at home, what was needed during past hospital and emergency department visits to treat pain and doses that have been effective & safe in the past.
  Patient-Specific Protocol: Patients assigned to this arm will be given pain medicine(s) based on pain medicine(s) they take at home and what was needed during their past hospital and emergency department visits to treat pain. Medicines include opioids, either morphine or hydromorphone. An outpatient SCD provider team will review patient's medical record to determine: 1) the patient's maximum home opioid dose, and 2) previous ED analgesic medication(s) and doses that have been effective & safe in the past. The patient's regular hematologist/sickle cell team will write the treatment plans. Medications will be given every 20-30 minutes for up to 6 hours.
  Morphine: 4 mg for participants weighing <50 kgs, 6mg for participants weighing 50-69.9 kgs, 8mg for participants weighing 70 - 89.9 kgs and 10mg for participants weighing greater than or equal to 90 kgs. dose is given. Re-dosing is every 20-30 minutes up to 6 hours with one possible dose escalation of 25%.
  Hydromorphone: 1 mg for participants weighing <60 kgs, 1.5 mg for participants weighing 60 - 89.9 kgs, and 2 mg for participants weighing greater than or equal to 90 kgs. dose is given. Re-dosing is every 20-30 minutes up to 6 hours with one possible dose escalation of 25%.
Period: Overall Study
Arm/Group | Patient-Specific Protocol | Weight-based Protocol
Started | 162 | 166
Completed | 50 | 46
Not Completed | 112 | 120
Not completed — No emergency department visit | 65 | 71
Not completed — Missed emergency department visit | 25 | 30
Not completed — Emergency Department visit for non vaso-occlusive episode diagnosis | 18 | 15
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — missing pain score | 1 | 1
Not completed — Confirmed COVID-19 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Participants arrived at the emergency department and once determined that they were not COVID + and were there for a vaso-occlusive episode and bed placement occurred, baseline data were collected. Baseline data were not collected on 8 participants following bed placement. 1 withdrew consent, 2 were investigator decision, 3 confirmed COVID + and 1 did not provide baseline information.
Groups:
- Patient-Specific Protocol: Patients assigned to this arm will be given pain medicine(s) based on pain medicine(s) they take at home and what was needed during their past hospital and emergency department visits to treat pain. Medicines include opioids, either morphine or hydromorphone. An outpatient SCD provider team will review patient's medical record to determine: 1) the patient's maximum home opioid dose, and 2) previous ED analgesic medication(s) and doses that have been effective & safe in the past. The patient's regular hematologist/sickle cell team will write the treatment plans. Medications will be given every 20-30 minutes for up to 6 hours.
  Morphine: 4 mg for participants weighing <50 kgs, 6mg for participants weighing 50-69.9 kgs, 8mg for participants weighing 70 - 89.9 kgs and 10mg for participants weighing greater than or equal to 90 kgs. dose is given. Re-dosing is every 20-30 minutes up to 6 hours with one possible dose escalation of 25%.
  Hydromorphone: 1 mg for participants weighing <60 kgs, 1.5 mg for participants weighing 60 - 89.9 kgs, and 2 mg for participants weighing greater than or equal to 90 kgs. dose is given. Re-dosing is every 20-30 minutes up to 6 hours with one possible dose escalation of 25%.
- Total: Total of all reporting groups
Arm/Group | Patient-Specific Protocol | Weight-based Protocol | Total
Number analyzed (Participants) | 54 | 50 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 50 | 104
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.3 (8.63) | 29.3 (8.28) | 30.3 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not collected on 1 participant
  Participants
    number analyzed (Participants) | 54 | 49 | 103
    Female | 36 | 28 | 64
    Male | 18 | 21 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected on 1 participant
  Participants
    number analyzed (Participants) | 54 | 49 | 103
    Hispanic or Latino | 2 | 0 | 2
    Not Hispanic or Latino | 52 | 49 | 101
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected on 1 participant
  Participants
    number analyzed (Participants) | 54 | 49 | 103
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 53 | 48 | 101
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54 | 50 | 104
Clinical Genotypes [Count of Participants; unit: Participants]
  SS, SB | 42 | 35 | 77
  SC SB+ | 12 | 15 | 27
Weight [Mean (Standard Deviation); unit: kg] | 73.8 (16.63) | 74.2 (16.49) | 74.0 (16.49)
Leg Ulcers [Count of Participants; unit: Participants] — Population: Data not collected on 1 participant
  Participants
    number analyzed (Participants) | 53 | 50 | 103
    (all) | 3 | 2 | 5
Pulmonary Hypertension [Count of Participants; unit: Participants] — Population: Data not collected on 3 participants
  Participants
    number analyzed (Participants) | 51 | 50 | 101
    (all) | 10 | 6 | 16
Acute Chest Syndrome [Count of Participants; unit: Participants] — Population: Data not collected on 3 participants
  Participants
    number analyzed (Participants) | 53 | 48 | 101
    (all) | 39 | 35 | 74
Retinopathy [Count of Participants; unit: Participants] — Population: Data not collected on 2 participants
  Participants
    number analyzed (Participants) | 53 | 49 | 102
    (all) | 2 | 4 | 6
Stroke [Count of Participants; unit: Participants] — Population: Data not collected on 4 participants
  Participants
    number analyzed (Participants) | 50 | 50 | 100
    (all) | 11 | 8 | 19
Transient ischemic attack [Count of Participants; unit: Participants] — Population: Data not collected on 6 participants
  Participants
    number analyzed (Participants) | 49 | 49 | 98
    (all) | 3 | 1 | 4
Avascular necrosis [Count of Participants; unit: Participants] — Population: Data not collected on 4 participants
  Participants
    number analyzed (Participants) | 53 | 47 | 100
    (all) | 22 | 17 | 39
Kidney dysfunction [Count of Participants; unit: Participants] — Population: Data not collected on 3 participants
  Participants
    number analyzed (Participants) | 51 | 50 | 101
    (all) | 2 | 5 | 7
Heart Failure [Count of Participants; unit: Participants] — Population: Data not collected on 2 participants
  Participants
    number analyzed (Participants) | 52 | 50 | 102
    (all) | 3 | 1 | 4
Gallbladder disease [Count of Participants; unit: Participants] — Population: Data not collected on 2 participants
  Participants
    number analyzed (Participants) | 52 | 50 | 102
    (all) | 18 | 15 | 33
Seizure [Count of Participants; unit: Participants] — Population: Data not collected on 4 participants
  Participants
    number analyzed (Participants) | 50 | 50 | 100
    (all) | 8 | 4 | 12
Liver Dysfunction [Count of Participants; unit: Participants] — Population: Data not collected on 2 participants
  Participants
    number analyzed (Participants) | 52 | 50 | 102
    (all) | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Change in Pain Score
Description: Pain is measured by having the patient mark pain on a scale of 0 to 100, with 0 being no pain and 100 being the worst pain ever. Pain scores were initially measured using a 0-100 millimeter visual analog scale with higher (closer to 100 being worse); however during the COVID-19 pandemic, one site removed paper forms from the emergency department as an infection control measure. The protocol was amended to add collection of a 0-100 verbal numerical rating scale and sites were ask to obtain both a vision and verbal score if possible collecting the visual score first. For the analysis, the visual score was used if available for the primary outcome. if not available, the verbal score was used.
Time Frame: baseline (bed placement), to disposition decision or a maximum treatment duration of 6 hours, whichever came first
Population: 3 participants were excluded following COVID-19 diagnosis, 5 participants had missing data following baseline so analysis could not be made.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient-Specific Protocol | Weight-based Protocol
Number analyzed (Participants) | 50 | 46
score on a scale | -27.0 (27.54) | -27.6 (28.13)
Statistical Analysis 1: Comparison: Patient-Specific Protocol vs Weight-based Protocol; Test type: Superiority; p = 0.909, Regression, Linear

2. Secondary Outcome: Length of Index ED (Emergency Department) Stay
Description: Length of index ED stay in hours from bed placement to discharge
Time Frame: From bed placement to discharge or 6 hours whichever comes first
Population: Patients had to be placed in bed in emergency department. Time was calculated from placement to change in disposition or at the end of 6 hours whichever came first.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Patient-Specific Protocol | Weight-based Protocol
Number analyzed (Participants) | 50 | 46
hours | 3.4 (1.48) | 4.2 (1.72)

3. Secondary Outcome: Length of Care
Description: Length of care from bed placement to last drug dose in hours.
Time Frame: up to 6 hours
Population: Data not collected on 10 participants
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Patient-Specific Protocol | Weight-based Protocol
Number analyzed (Participants) | 49 | 45
hours | 2.5 (1.46) | 2.6 (1.62)

4. Secondary Outcome: Total Number of Hospitalizations for Vaso-Occlusive Episode 7 Days Post Enrollment
Description: Number of hospitalizations for Vaso-Occlusive Episode (VOE) within 7 days following enrollment
Time Frame: Up to 7 days post enrollment
Measure: Number; unit: hospitalizations
Arm/Group | Patient-Specific Protocol | Weight-based Protocol
Number analyzed (Participants) | 50 | 46
hospitalizations | 11 | 14

5. Secondary Outcome: Number of Participants Experiencing Side Effects
Description: Side effects and safety at any time during the emergency department visit
Time Frame: Bed placement to discharge or 6 hours, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Patient-Specific Protocol | Weight-based Protocol
Number analyzed (Participants) | 50 | 46
Participants
  Nausea | 19 | 19
  vomiting | 7 | 6
  pruritus | 31 | 36
  SPO2<95% requiring supplemental oxygen via nasal cannula due to opioid therapy | 4 | 7
  Moderate to severe sedation (sedation score of >=3 | 4 | 5
  Drowsiness | 15 | 9
  respiratory depression not requiring intubation | 0 | 1
  Low blood pressure (SBP,90mmHg and/or DBP<50mmHg | 3 | 1

ADVERSE EVENTS:
Time Frame: From enrollment in the emergency department through 7 days post enrollment for up to 8 days.
Groups:
- Patient-Specific Protocol: Patients assigned to this treatment protocol will be given pain medicine(s) based on pain medicine(s) taken at home & what was needed during past emergency department visits to treat pain. Medicines include opioids, morphine or hydromorphone. A member of the outpatient provider team reviews patient's medical record to determine patient's maximum home opioid dose, previous ED analgesic medication(s) & doses that have been effective & safe in the past. Patient's regular hematologist/sickle cell team will write the treatment plans.
  Medications will be given every 20-30 minutes for up to 6 hours. Morphine: 4 mg for participants weighing <50 kgs, 6mg for participants weighing 50-69.9 kgs, 8mg for participants weighing 70 - 89.9 kgs and 10mg for participants weighing > or equal to 90 kgs. Re-dosing is every 20-30 minutes up to 6 hours with one possible dose escalation of 25%.
  Hydromorphone: 1 mg for participants weighing <60 kgs, 1.5 mg for participants weighing 60 - 89.9 kgs, and 2 mg for participants weighing > or equal to 90 kgs. Re-dosing is every 20-30 minutes up to 6 hours with one possible dose escalation of 25%.
  There are only two, not four, randomized interventions in this trial: patient specific pain management protocol and weight-based pain management protocol. Here the word "protocol" refers to pain management approach. The AEs have been submitted by each of these two interventions.
- Weight-based Protocol: Patients assigned to this treatment protocol will be given pain medicine(s) based on their weight.
  Weight-based Protocol: Patients assigned to this treatment protocol will be given pain medicine(s) based on their weight. Medicines will include opioids, either morphine or hydromorphone. Plans will be written by the patients regular hematologist/sickle cell team.
  Morphine: 4 mg for participants weighing <50 kgs, 6mg for participants weighing 50-69.9 kgs, 8mg for participants weighing 70 - 89.9 kgs and 10mg for participants weighing greater than or equal to 90 kgs. dose is given. Re-dosing is every 20-30 minutes up to 6 hours with one possible dose escalation of 25%.
  Hydromorphone: 1 mg for participants weighing <60 kgs, 1.5 mg for participants weighing 60 - 89.9 kgs, and 2 mg for participants weighing greater than or equal to 90 kgs. dose is given. Re-dosing is every 20-30 minutes up to 6 hours with one possible dose escalation of 25%.
  There are only two, not four, randomized interventions in this trial: patient specific pain management protocol and weight-based pain management protocol. Here the word "protocol" refers to pain management approach. The AEs have been submitted by each of these two interventions.
Arm/Group | Patient-Specific Protocol | Weight-based Protocol
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/46
Other Adverse Events (participants affected / at risk) | 50/50 | 46/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient-Specific Protocol (N=50) | Weight-based Protocol (N=46)
nausea (General disorders) | 19 (19) | 19 (19)
vomiting (General disorders) | 7 (7) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 31 (31) | 36 (36)
SPO2<95% (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)
Moderate to severe sedation (General disorders) | 4 (4) | 5 (5)
Drowsiness (General disorders) | 15 (15) | 9 (9)
Respiratory depression not requiring intubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
low blood pressure (General disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT03933397/Prot_001.pdf
  • Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT03933397/SAP_003.pdf
  • Informed Consent Form (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT03933397/ICF_000.pdf